CLINICAL TRIAL: NCT03459612
Title: A Phase I, Randomized, Subject- and Investigator-Blind, Placebo-Controlled, 4-Period Cross-Over Study Assessing the Duration of Effect of Lasmiditan on Simulated Driving Performance in Healthy Volunteers
Brief Title: A Study of Lasmiditan on Simulated Driving Performance in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 17048; H8H-MC-LAIF (Other: Eli Lilly and Company)
Record Dates: First submitted 2018-03-02; First posted 2018-03-09 (Actual); Results first posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2019-12

CONDITIONS: Healthy
MeSH Terms: interventions — lasmiditan; Diphenhydramine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Placebo administered orally in one of four study periods.
  Interventions: Drug: Placebo
- 100 milligrams (mg) Lasmiditan (Experimental): 100 mg lasmiditan administered orally in one of four study periods.
  Interventions: Drug: Lasmiditan
- 200 mg Lasmiditan (Experimental): 200 mg lasmiditan administered orally in one of four study periods.
  Interventions: Drug: Lasmiditan
- Diphenhydramine (Active Comparator): 50 mg diphenhydramine administered orally in one of four study periods.
  Interventions: Drug: Diphenhydramine

INTERVENTIONS:
Drug: Lasmiditan — Administered orally
  Other Names: LY573144
  Arms: 100 milligrams (mg) Lasmiditan; 200 mg Lasmiditan
Drug: Placebo — Administered orally
  Arms: Placebo
Drug: Diphenhydramine — Administered orally
  Arms: Diphenhydramine

SUMMARY:
The purpose of this study is to evaluate the effect of lasmiditan on simulated driving performance in healthy participants. Participants are expected to complete each of four study periods, which will last a total of about 10 days. During this time, participants will remain in the clinical research unit. Screening must be completed within 28 days before the start of the study. Follow-up will be completed about one week after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy males or females, as determined through medical history and physical examination.
* Possess a valid driver's license and is an active driver at screening. Driven a minimum of 8,000 miles (about 13,000 kilometers) per year for the preceding 3 years.
* Have a score of <10 on the Epworth Sleepiness Scale.

Exclusion Criteria:

* Have a history within 3 months of admission, or current treatment for, a sleeping disorder (including excessive snoring, obstructive sleep apnea), or a chronic painful condition that interferes with the subject's sleep.
* Have a history of difficulty either falling asleep or staying asleep in the previous 3 months of admission that is considered clinically significant by the investigator.
* Are expected to use any other medication or dietary supplement to promote sleep including over the-counter sleep medications, during their participation in the study.
* Have traveled across 2 or more time zones (transmeridian travel) in the past 2 weeks prior to randomization.
* Have worked in a night shift in the past 2 weeks prior to randomization.
* Show a history of central nervous system (CNS) conditions such as strokes, transient ischemic attacks, significant head trauma, seizures, CNS infections, migraine, brain surgery, or any other neurological conditions that, in the opinion of the investigator, increase the risk of participating in the study.
* Show evidence of significant active neuropsychiatric disease (e.g., manic depressive illness, schizophrenia, depression) considered as clinically significant by the investigator.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2018-03-26 (Actual); Primary Completion 2018-06-23 (Actual); Study Completion 2018-06-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- United States (3):
  - Covance Clinical Research Inc, Daytona Beach, Florida
  - Covance, Dallas, Texas
  - Covance Clinical Research Inc, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Randomized, 4-period cross-over study in healthy participants.
Groups:
- Sequence 1: Period 1: Placebo administered PO. Period 2: 100 mg lasmiditan administered PO. Period 3: 50 mg diphenhydramine administered PO. Period 4: 200 mg lasmiditan administered PO. Study treatments were administered at up to 4 dosing occasions (0, 6, and 10 hours on Day 1 and 22 hours on Day 2) within each period: lasmiditan was only administered at 0 hours.
  Each period is 3 days duration
- Sequence 2: Period 1: 100 mg lasmiditan administered PO. Period 2: 200 mg lasmiditan administered PO. Period 3: Placebo administered PO. Period 4: 50 mg diphenhydramine administered PO. Study treatments were administered at up to 4 dosing occasions (0, 6, and 10 hours on Day 1 and 22 hours on Day 2) within each period: lasmiditan was only administered at 0 hours. Each period is 3 days duration
- Sequence 3: Period 1: 200 mg lasmiditan administered PO Period 2 : 50 mg diphenhydramine administered PO Period 3: 100 mg lasmiditan administered PO Period 4: Placebo administered PO Study treatments were administered at up to 4 dosing occasions (0, 6, and 10 hours on Day 1 and 22 hours on Day 2) within each period: lasmiditan was only administered at 0 hours.
  Each period is 3 days duration
- Sequence 4: Period 1: 50 mg diphenhydramine administered PO Period 2: Placebo administered PO Period 3: 200 mg lasmiditan administered PO Period 4: 100 mg lasmiditan administered PO Study treatments were administered at up to 4 dosing occasions (0, 6, and 10 hours on Day 1 and 22 hours on Day 2) within each period: lasmiditan was only administered at 0 hours.
  Each period is 3 days duration
Period: Period 1
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 17 | 17 | 17 | 17
Received at Least 1 Dose of Study Drug | 17 | 17 | 17 | 17
Completed | 17 | 17 | 17 | 17
Not Completed | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 17 | 17 | 17 | 17
Received at Least 1 Dose of Study Drug | 17 | 17 | 17 | 17
Completed | 17 | 17 | 17 | 17
Not Completed | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 17 | 17 | 17 | 17
Received at Least 1 Dose of Study Drug | 17 | 17 | 17 | 17
Completed | 17 | 17 | 17 | 17
Not Completed | 0 | 0 | 0 | 0
Period: Period 4
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 17 | 17 | 16 (One participant completed period 3 and withdrew for personal reasons prior to Period 4.) | 17
Received at Least 1 Dose of Study Drug | 17 | 17 | 16 | 17
Completed | 17 | 17 | 16 | 17
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least 1 dose of study drug.
Groups:
- Sequence 1: Participants received Placebo, 100 mg lasmiditan, 200 mg lasmiditan, 50 mg diphenhydramine as per below sequence.
  Period 1: Placebo administered PO. Period 2: 100 mg lasmiditan administered PO. Period 3: 50 mg diphenhydramine administered PO. Period 4: 200 mg lasmiditan administered PO. Study treatments were administered at up to 4 dosing occasions (0, 6, and 10 hours on Day 1 and 22 hours on Day 2) within each period: lasmiditan was only administered at 0 hours.
  Each period is 3 days duration
- Sequence 2: Participants received Placebo, 100 mg lasmiditan, 200 mg lasmiditan, 50 mg diphenhydramine as per below sequence.
  Period 1: 100 mg lasmiditan administered PO. Period 2: 200 mg lasmiditan administered PO. Period 3: Placebo administered PO. Period 4: 50 mg diphenhydramine administered PO. Study treatments were administered at up to 4 dosing occasions (0, 6, and 10 hours on Day 1 and 22 hours on Day 2) within each period: lasmiditan was only administered at 0 hours.
  Each period is 3 days duration
- Sequence 3: Participants received Placebo, 100 mg lasmiditan, 200 mg lasmiditan, 50 mg diphenhydramine as per below sequence.
  Period 1: 200 mg lasmiditan administered PO Period 2 : 50 mg diphenhydramine administered PO Period 3: 100 mg lasmiditan administered PO Period 4: Placebo administered PO Study treatments were administered at up to 4 dosing occasions (0, 6, and 10 hours on Day 1 and 22 hours on Day 2) within each period: lasmiditan was only administered at 0 hours.
  Each period is 3 days duration
- Sequence 4: Participants received Placebo, 100 mg lasmiditan, 200 mg lasmiditan, 50 mg diphenhydramine as per below sequence.
  Period 1: 50 mg diphenhydramine administered PO Period 2: Placebo administered PO Period 3: 200 mg lasmiditan administered PO Period 4: 100 mg lasmiditan administered PO Study treatments were administered at up to 4 dosing occasions (0, 6, and 10 hours on Day 1 and 22 hours on Day 2) within each period: lasmiditan was only administered at 0 hours.
  Each period is 3 days duration
- Total: Total of all reporting groups
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Total
Number analyzed (Participants) | 17 | 17 | 17 | 17 | 68
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 17 | 17 | 17 | 17 | 68
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 6 | 10 | 28
  Male | 10 | 12 | 11 | 7 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 6 | 1 | 12
  Not Hispanic or Latino | 13 | 16 | 11 | 16 | 56
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 2 | 1 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 7 | 5 | 3 | 4 | 19
  White | 9 | 9 | 11 | 12 | 41
  More than one race | 0 | 1 | 2 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17 | 17 | 17 | 17 | 68

OUTCOME MEASURES:

1. Primary Outcome: Simulated Driving Performance in Healthy Participants as Measured by Standard Deviation of Lateral Position (SDLP) Using the Cognitive Research Corporation Driving Simulator-MiniSim (CRCDS-MiniSim)
Description: The standard deviation of lateral position (SDLP) is the primary parameter used as stable measure of driving performance with high test-retest reliability. It measures the driver's ability to stay in a constant position within the driving lane.
  LS Means were analyzed using a mixed repeated measures model with fixed effects for sequence, period, and treatment, with repeated observations for subjects for each of the driving time points.
Time Frame: 8 hours postdose in each dosing period
Population: All randomized participants who received at least 1 dose of study drug and had evaluable data.
Measure: Least Squares Mean (Full Range); unit: centimeters
Groups:
- 100 mg Lasmiditan: 100 milligrams (mg) Lasmiditan administered orally (PO) in one of four study periods.
- 200 mg Lasmiditan: 200 mg Lasmiditan administered PO in one of four study periods.
- 50 mg Diphenhydramine: Diphenhydramine administered PO in one of four study periods.
Arm/Group | Placebo | 100 mg Lasmiditan | 200 mg Lasmiditan | 50 mg Diphenhydramine
Number analyzed (Participants) | 67 | 68 | 68 | 68
centimeters | 29.85 [19.7 to 49.0] | 30.83 [18.9 to 52.7] | 31.61 [21.6 to 49.3] | 34.83 [19.2 to 62.5]
Statistical Analysis 1: Comparison: Placebo vs 100 mg Lasmiditan; Test type: Non-Inferiority — Non-inferiority p-value tests null hypothesis that difference in LS means ≥ 4.4 versus alternative hypothesis that difference in Least Square (LS) means < 4.4; p < 0.0001, Mixed Models Analysis; Difference in LS Means = 0.98, 95% CI 2-sided [-0.43 to 2.39]
Statistical Analysis 2: Comparison: Placebo vs 200 mg Lasmiditan; Test type: Non-Inferiority — Non-inferiority p-value tests null hypothesis that difference in LS means ≥ 4.4 versus alternative hypothesis that difference in LS means < 4.4; p < 0.0001, Mixed Models Analysis; LS Means = 1.76, 95% CI 2-sided [0.32 to 3.20]
Statistical Analysis 3: Comparison: Placebo vs 50 mg Diphenhydramine; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; p < 0.0001, Mixed Models Analysis; LS Means = 4.98, 95% CI 2-sided [3.58 to 6.38]

2. Primary Outcome: Simulated Driving Performance in Healthy Participants as Measured by Standard Deviation of Lateral Position (SDLP) Using the Cognitive Research Corporation Driving Simulator-MiniSim (CRCDS-MiniSim)
Description: as for outcome 1
Time Frame: 12 hours postdose in each dose period
Population: All randomized participants who received at least 1 dose of study drug and had evaluable data.
Measure: Least Squares Mean (Full Range); unit: centimeters
Groups:
- Placebo: Placebo administered orally (PO) in one of four study periods.
Arm/Group | Placebo | 100 mg Lasmiditan | 200 mg Lasmiditan | 50 mg Diphenhydramine
Number analyzed (Participants) | 67 | 67 | 68 | 68
centimeters | 30.41 [18.4 to 54.6] | 30.29 [19.1 to 50.4] | 30.09 [19.9 to 48.6] | 34.72 [19.7 to 56.2]
Statistical Analysis 1: Comparison: Placebo vs 100 mg Lasmiditan; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; p < 0.0001, Mixed Models Analysis; Difference in LS Means = -0.12, 95% CI 2-sided [-1.28 to 1.04]
Statistical Analysis 2: Comparison: Placebo vs 200 mg Lasmiditan; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; p < 0.0001, Mixed Models Analysis; Difference in LS Means = -0.32, 95% CI 2-sided [-1.51 to 0.88]
Statistical Analysis 3: Comparison: Placebo vs 50 mg Diphenhydramine; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; p < 0.0001, Mixed Models Analysis; Difference in LS Means = 4.31, 95% CI 2-sided [3.17 to 5.45]

3. Primary Outcome: Simulated Driving Performance in Healthy Participants as Measured by Standard Deviation of Lateral Position (SDLP) Using the Cognitive Research Corporation Driving Simulator-MiniSim (CRCDS-MiniSim)
Description: as for outcome 1
Time Frame: 24 hours post dose in each dose period
Population: All randomized participants who received at least 1 dose of study drug and had evaluable data.
Measure: Least Squares Mean (Full Range); unit: centimeters
Arm/Group | Placebo | 100 mg Lasmiditan | 200 mg Lasmiditan | 50 mg Diphenhydramine
Number analyzed (Participants) | 67 | 68 | 68 | 68
centimeters | 32.04 [18.5 to 57.5] | 31.07 [18.6 to 54.8] | 31.00 [19.9 to 55.7] | 36.10 [19.3 to 66.7]
Statistical Analysis 1: Comparison: Placebo vs 100 mg Lasmiditan; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; p < 0.0001, Mixed Models Analysis; Differnce in LS Means = -0.97, 95% CI 2-sided [-2.30 to 0.36]
Statistical Analysis 2: Comparison: Placebo vs 200 mg Lasmiditan; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; p < 0.0001, Mixed Models Analysis; Difference in LS Means = -1.04, 95% CI 2-sided [-2.40 to 0.32]
Statistical Analysis 3: Comparison: Placebo vs 50 mg Diphenhydramine; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; p < 0.0001, Mixed Models Analysis; Difference in LS Means = 4.05, 95% CI 2-sided [2.73 to 5.38]

4. Secondary Outcome: Karolinska Sleepiness Scale (KSS) Score
Description: The KSS is used to assess subjective level of sleepiness. This is a participant self-report measure of situational sleepiness and provides an assessment of alertness/sleepiness at a particular point in time. It is a 9-point categorical Likert scale on which the participant rates sleepiness from 1 (very alert) to 9 (very sleepy/fighting sleep), with higher scores indicating more sleepiness and lower scores indicating more alertness.
Time Frame: 8 hours postdose in each dose period
Population: All randomized participant that received at least 1 dose of study drug and had evaluable data.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | 100 mg Lasmiditan | 200 mg Lasmiditan | 50 mg Diphenhydramine
Number analyzed (Participants) | 67 | 68 | 68 | 68
Units on a scale | 3.19 (1.61) | 3.46 (1.65) | 3.90 (1.78) | 3.93 (1.76)
Statistical Analysis 1: Comparison: Placebo vs 100 mg Lasmiditan; Test type: Superiority; Differences of Least Square Mean = 0.28, 95% CI 2-sided [-0.15 to 0.70]
Statistical Analysis 2: Comparison: Placebo vs 200 mg Lasmiditan; Test type: Superiority; Difference of Least Square Means = 0.66, 95% CI 2-sided [0.22 to 1.10]
Statistical Analysis 3: Comparison: Placebo vs 50 mg Diphenhydramine; Test type: Superiority; Difference of Least Square Means = 0.81, 95% CI 2-sided [0.39 to 1.24]

5. Secondary Outcome: Karolinska Sleepiness Scale (KSS) Score
Description: as for outcome 4
Time Frame: 12 hours postdose in each dose period
Population: All randomized participants who received at least 1 dose of study drug and had evaluable data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | 100 mg Lasmiditan | 200 mg Lasmiditan | 50 mg Diphenhydramine
Number analyzed (Participants) | 67 | 68 | 67 | 68
units on a scale | 3.43 (1.57) | 3.94 (1.62) | 3.79 (1.74) | 4.74 (2.05)
Statistical Analysis 1: Comparison: Placebo vs 100 mg Lasmiditan; Test type: Superiority; Difference of Least Square Means = 0.48, 95% CI 2-sided [0.00 to 0.96]
Statistical Analysis 2: Comparison: Placebo vs 200 mg Lasmiditan; Test type: Superiority; Differnce of Least Square Means = 0.34, 95% CI 2-sided [-0.14 to 0.82]
Statistical Analysis 3: Comparison: Placebo vs 50 mg Diphenhydramine; Test type: Superiority; Difference of Least Square Means = 1.29, 95% CI 2-sided [0.81 to 1.78]

6. Secondary Outcome: Karolinska Sleepiness Scale (KSS) Score
Description: as for outcome 4
Time Frame: 24 hours postdose in each dose period
Population: All randomized participants that received at least 1 dose of study drug and had evaluable data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | 100 mg Lasmiditan | 200 mg Lasmiditan | 50 mg Diphenhydramine
Number analyzed (Participants) | 67 | 68 | 68 | 67
units on a scale | 4.19 (2.02) | 3.72 (1.69) | 3.93 (2.13) | 4.75 (2.15)
Statistical Analysis 1: Comparison: Placebo vs 200 mg Lasmiditan; Test type: Superiority; Difference of Least Square Means = -0.58, 95% CI 2-sided [-1.10 to -0.06]
Statistical Analysis 2: Comparison: Placebo vs 200 mg Lasmiditan; Test type: Superiority; Difference of Least Square Means = -0.40, 95% CI 2-sided [-0.89 to 0.09]
Statistical Analysis 3: Comparison: Placebo vs 50 mg Diphenhydramine; Test type: Superiority; Difference of Least Square Means = 0.44, 95% CI 2-sided [-0.09 to 0.96]

7. Secondary Outcome: Number of Correct Responses in Driving Performance Using CogScreen Symbol Digit Coding (SDC) Test
Description: The SDC Test, a digit symbol substitution test that is sensitive to changes in information processing speed, provides measures of response speed and accuracy. The test was administered prior to the simulated driving sessions. The principal test score measures the number of correct responses in 120 seconds. SDC was used in this study to measure attention, visual scanning, working memory, and speed of information processing. A measure of recall accuracy A higher score indicates greater processing speed
Time Frame: 8 hours postdose in each dose period
Population: All randomized participant that received at least 1 dose of study drug and had evaluable data.
Measure: Mean (Standard Deviation); unit: Correct responses
Arm/Group | Placebo | 100 mg Lasmiditan | 200 mg Lasmiditan | 50 mg Diphenhydramine
Number analyzed (Participants) | 67 | 67 | 67 | 68
Correct responses | 69.48 (11.32) | 69.76 (10.17) | 68.88 (11.27) | 69.01 (11.21)
Statistical Analysis 1: Comparison: Placebo vs 100 mg Lasmiditan; Test type: Superiority; Difference in Least Square Means = 0.00, 95% CI 2-sided [-1.61 to 1.62]
Statistical Analysis 2: Comparison: Placebo vs 200 mg Lasmiditan; Test type: Superiority; Difference in Lease Square Means = -0.74, 95% CI 2-sided [-2.49 to 1.01]
Statistical Analysis 3: Comparison: Placebo vs 50 mg Diphenhydramine; Test type: Superiority; Difference in Least Square Means = -0.72, 95% CI 2-sided [-2.32 to 0.89]

8. Secondary Outcome: Number of Correct Responses in Driving Performance Using CogScreen Symbol Digit Coding (SDC) Test
Description: The SDC Test, a digit symbol substitution test that is sensitive to changes in information processing speed, provides measures of response speed and accuracy. The test was administered prior to the simulated driving sessions. The principal test score measures the number of correct responses in 120 seconds. SDC was used in this study to measure attention, visual scanning, working memory, and speed of information processing. Scores range from 0 (No correct responses). A higher score indicates greater processing speed.
Time Frame: 12 hours postdose in each dose period
Population: All randomized participants who received study drug and have evaluable data.
Measure: Mean (Standard Deviation); unit: Correct responses
Arm/Group | Placebo | 100 mg Lasmiditan | 200 mg Lasmiditan | 50 mg Diphenhydramine
Number analyzed (Participants) | 67 | 68 | 68 | 68
Correct responses | 71.33 (11.26) | 70.91 (9.87) | 72.16 (9.91) | 68.21 (10.04)
Statistical Analysis 1: Comparison: Placebo vs 100 mg Lasmiditan; Test type: Superiority; Difference of Least Square Means = -1.79, 95% CI 2-sided [-3.52 to -0.06]
Statistical Analysis 2: Comparison: Placebo vs 200 mg Lasmiditan; Test type: Superiority; Difference in Least Square Means = -0.29, 95% CI 2-sided [-2.00 to 1.42]
Statistical Analysis 3: Comparison: Placebo vs 50 mg Diphenhydramine; Test type: Superiority; Difference in Least Square Means = -3.81, 95% CI 2-sided [-5.53 to -2.08]

9. Secondary Outcome: Number of Correct Responses in Driving Performance Using CogScreen Symbol Digit Coding (SDC) Test
Description: as for outcome 8
Time Frame: 24 hours postdose in each dose period
Population: All randomized participants who received study drug and have evaluable data.
Measure: Mean (Standard Deviation); unit: Correct responses
Arm/Group | Placebo | 100 mg Lasmiditan | 200 mg Lasmiditan | 50 mg Diphenhydramine
Number analyzed (Participants) | 67 | 68 | 68 | 68
Correct responses | 70.78 (9.84) | 70.53 (10.52) | 70.66 (10.24) | 68.31 (10.27)
Statistical Analysis 1: Comparison: Placebo vs 100 mg Lasmiditan; Test type: Superiority; Difference of Least Square Means = -0.28, 95% CI 2-sided [-1.71 to 1.15]
Statistical Analysis 2: Comparison: Placebo vs 200 mg Lasmiditan; Test type: Superiority; Difference of Least Square Means = -0.31, 95% CI 2-sided [-1.71 to 1.08]
Statistical Analysis 3: Comparison: Placebo vs 50 mg Diphenhydramine; Test type: Superiority; Difference of Least Square Means = -2.70, 95% CI 2-sided [-4.13 to -1.27]

10. Secondary Outcome: Total Number of Collisions
Description: Total collisions are the sum off collisions with other vehicles and off-road crashes. Collision counts also included the number of times that a lane deviation exceeded 4 feet but where no collision occurred ( a crash-likely event).
Time Frame: 8 hours postdose in each dose period
Population: All randomized participants who received at least 1 dose of study drug and had evaluable data.
Measure: Mean (Standard Deviation); unit: collisions
Arm/Group | Placebo | 100 mg Lasmiditan | 200 mg Lasmiditan | 50 mg Diphenhydramine
Number analyzed (Participants) | 67 | 68 | 68 | 68
collisions | 0.1 (0.2) | 0.0 (0.2) | 0.0 (0.1) | 0.4 (1.1)
Statistical Analysis 1: Comparison: Placebo vs 100 mg Lasmiditan; Test type: Superiority; p = 0.6875, Wilcoxon Signed Rank test; Mean Difference (Final Values) = -0.03, Standard Deviation 0.30
Statistical Analysis 2: Comparison: Placebo vs 200 mg Lasmiditan; Test type: Superiority; p = 0.3750, Wilcoxon Signed Rank test; Mean Difference (Final Values) = -0.04, Standard Deviation 0.27
Statistical Analysis 3: Comparison: Placebo vs 50 mg Diphenhydramine; Test type: Superiority; p = 0.0115, Wilcoxon Signed Rank test; Mean Difference (Final Values) = 0.30, Standard Deviation 1.00

11. Secondary Outcome: Total Number of Collisions
Description: as for outcome 10
Time Frame: 12 hours postdose in each dose period
Population: All randomized participants who received at least 1 dose of study drug and had evaluable data.
Measure: Mean (Standard Deviation); unit: collisions
Arm/Group | Placebo | 100 mg Lasmiditan | 200 mg Lasmiditan | 50 mg Diphenhydramine
Number analyzed (Participants) | 67 | 67 | 68 | 68
collisions | 0.1 (0.4) | 0.0 (0.1) | 0.1 (0.3) | 0.2 (0.7)
Statistical Analysis 1: Comparison: Placebo vs 100 mg Lasmiditan; Test type: Superiority; p = 0.1563, Wilcoxon Signed Rank test; Mean Difference (Final Values) = -0.09, Standard Deviation 0.42
Statistical Analysis 2: Comparison: Placebo vs 200 mg Lasmiditan; Test type: Superiority; p = 0.5938, Wilcoxon Signed Rank test; Mean Difference (Final Values) = -0.04, Standard Deviation 0.44
Statistical Analysis 3: Comparison: Placebo vs 50 mg Diphenhydramine; Test type: Superiority; p = 0.0938, Wilcoxon Signed Rank test; Mean Difference (Final Values) = 0.12, Standard Deviation 0.54

12. Secondary Outcome: Total Number of Collisions
Description: as for outcome 10
Time Frame: 24 hours postdose in each dose period
Population: All randomized participants who received at least 1 dose of study drug and had evaluable data.
Measure: Mean (Standard Deviation); unit: collisions
Arm/Group | Placebo | 100 mg Lasmiditan | 200 mg Lasmiditan | 50 mg Diphenhydramine
Number analyzed (Participants) | 67 | 68 | 68 | 68
collisions | 0.2 (0.6) | 0.0 (0.2) | 0.2 (0.7) | 0.6 (1.7)
Statistical Analysis 1: Comparison: Placebo vs 100 mg Lasmiditan; Test type: Superiority; p = 0.1250, Wilcoxon Signed Rank test; Mean Difference (Final Values) = -0.12, Standard Deviation 0.56
Statistical Analysis 2: Comparison: Placebo vs 200 mg Lasmiditan; Test type: Superiority; p = 0.9590, Wilcoxon Signed Rank test; Mean Difference (Final Values) = 0.03, Standard Deviation 0.94
Statistical Analysis 3: Comparison: Placebo vs 50 mg Diphenhydramine; Test type: Superiority; p = 0.0097, Wilcoxon Signed Rank test; Mean Difference (Final Values) = 0.46, Standard Deviation 1.76

13. Secondary Outcome: Pharmacokinetics (PK): Maximum Observed Drug Concentration (Cmax) of Lasmiditan
Description: PK: Cmax of Lasmiditan
Time Frame: Day 1: Predose, 0.5 hour (hr), 1hr, 1.5hr, 2hr, 3hr, 4hr, 6hr, 8hr, 10 hr, 12hr, 24hr, 36hr, 48hr postdose
Population: All randomized participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter
Arm/Group | 100 mg Lasmiditan | 200 mg Lasmiditan
Number analyzed (Participants) | 68 | 67
nanograms per milliliter | 183 (31) | 366 (30)

14. Secondary Outcome: PK: Area Under the Concentration Versus Time Curve (AUC) of Lasmiditan to the Last Timepoint (0-tlast)
Description: PK: AUC of Lasmiditan until the last time a concentration is detected.
Time Frame: Day 1: Predose, 0.5 hour (hr), 1hr, 1.5hr, 2hr, 3hr, 4hr, 6hr, 8hr, 10 hr, 12hr, 24hr, 36hr, 48hr postdose
Population: All randomized participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hour per milliliter
Arm/Group | 100 mg Lasmiditan | 200 mg Lasmiditan
Number analyzed (Participants) | 67 | 67
ng*hour per milliliter | 1060 (28) | 2230 (25)

ADVERSE EVENTS:
Time Frame: up to 4 months
Description: All randomized participants who received at least 1 dose of study drug.
Arm/Group | Placebo | 100 mg Lasmiditan | 200 mg Lasmiditan | 50 mg Diphenhydramine
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/68 | 0/68 | 0/68
Serious Adverse Events (participants affected / at risk) | 0/67 | 0/68 | 0/68 | 0/68
Other Adverse Events (participants affected / at risk) | 6/67 | 23/68 | 25/68 | 7/68
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=67) | 100 mg Lasmiditan (N=68) | 200 mg Lasmiditan (N=68) | 50 mg Diphenhydramine (N=68)
Nausea (Gastrointestinal disorders) | 4 (4) | 2 (2) | 2 (2) | 1 (1)
Fatigue (General disorders) | 1 (1) | 6 (7) | 4 (4) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 11 (11) | 12 (12) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 3 (3) | 6 (6) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 4 (4) | 6 (6) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 5 (6) | 7 (7) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-02-21): https://cdn.clinicaltrials.gov/large-docs/12/NCT03459612/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-22): https://cdn.clinicaltrials.gov/large-docs/12/NCT03459612/SAP_001.pdf